CLINICAL TRIAL: NCT02314312
Title: A 12 Month, Single-center, Open-label, Randomized-controlled Trial to Investigate Efficacy, Safety and Tolerability of Everolimus in Combination With Cyclosporine A and Corticosteroid in de Novo Transplant Recipients of Expanded Criteria Donor Kidneys or Acute Kidney Injury
Brief Title: Efficacy and Safety of Everolimus in de Novo Kidney Transplant Recipients of ECD or AKI Donors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, CHALERMPON NA PETVICHARN, Ramathibodi Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ATH01T
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Transplantation of Kidney; Expanded Criteria Donor; ECD
Keywords: Kidney transplantation; ECD
MeSH Terms: interventions — Everolimus; Cyclosporine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: investigation arm (Experimental): De novo kidney transplantation form ECD/AKI donor with Everolimus + low dose cyclosporinA + prednisolone as immunosuppressive regimen
  Interventions: Drug: Everolimus + low dose cyclosporin A + prednisolone
- B: control arm (Other): De novo kidney transplantation form ECD/AKI donor with standard immunosuppressive regimen
  Interventions: Drug: Standard immunosupressive regimen

INTERVENTIONS:
Drug: Everolimus + low dose cyclosporin A + prednisolone
  Arms: A: investigation arm
Drug: Standard immunosupressive regimen
  Arms: B: control arm

SUMMARY:
Single center, open-label randomized-control trial Population: de novo 48 kidney transplant recipients (age 18-75 years) from ECD/AKI donors Compare: everolimus with low dose CNI and prednisolone versus standard immunosuppressive regimen Objective: To evaluate efficacy of everolimus with low dose CNI in de novo kidney transplant recipients of ECD/AKI donors Primary endpoint: Mean eGFR (CKD-EPI) at 12 months post-transplantation

DETAILED DESCRIPTION:
Secondary Endpoints:

* To assess renal function by means of eGFR (Cockcrault and Gault formula), at -Month 6 and 12 post-transplantation
* To assess incidence of the individual composite endpoints including BPAR, graft loss and death at Month 6 and 12 post-transplantation
* To assess the incidence and duration of renal replacement therapy
* To assess the incidence of chronic allograft nephropathy (IF/TA) at Month 12
* To assess renal function by means of serum creatinine at Month 6 and 12 post-transplantation
* To compare the overall safety and tolerability (incidence of AEs and SAEs, infections, discontinuations due to AEs, lab abnormalities, wound and surgical complications) at Month 6 and 12 post-transplantation

Definition of ECD

* Brain-dead donor > 60 years old or
* Donor age > 50 years old with two of the following criteria;
* History of HT
* Terminal SCr. ≥ 1.5 mg/dL
* Death from cerebrovascular accident Definition of AKI donor
* Brain-dead donor with an increase of SCr. ≥ 0.3 mg/dL from baseline

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Recipients of first DDKT from ECD or AKI donors
* Patient willing to participate in the study

Exclusion Criteria:

* Multi-organ recipients

  * Organ donation after Cardiac Death (DCD).
  * PRA > 20 % or with historical peak PRA > 50%
  * Patients who lost first graft due to immunological reason within the first year post-transplantation.
  * ABO incompatible transplants or positive cross-match
  * Patients with chronic inflammatory bowel disease.
  * Severe allergy requiring acute treatment, or any known hypersensitivity to everolimus, thymoglobulin
  * Thrombocytopenia (platelet < 75,000/mm3), ANC < 1,500 /mm3 or leucopenia (leucocytes < 2,500/mm3), or Hb < 6 g/dL
  * Chronic active HCV, HIV, or HBsAg positive
  * History of malignancy during the last five years, except squamous or basal cell carcinoma of the skin.
  * Ongoing infection requiring treatment with a systemic antibiotic.
  * Patient with severe hypercholesterolemia (> 300 mg/dL) or hypertriglyceridemia (> 600 mg/dL) that cannot be controlled
  * Evidence of severe liver disease.
  * Severe restrictive or obstructive pulmonary disorders.
  * Pregnant or nursing (lactating) women.
  * Patient who refuse to participate into the study or would like to withdraw from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
eGFR (CKD-EPI) | 12 months post kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Kantachuvesiri, M.D., PH.D, Principal Investigator — Ramathibodi Hospital, Mahidol University